CLINICAL TRIAL: NCT02931110
Title: A Phase 1 Dose-Escalation and Cohort-Expansion Study of Intravenous CBL0137 in Subjects With Previously Treated Hematological Cancers
Brief Title: Study of IV CBL0137 in Previously Treated Hematological Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Incuron (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: I137-102
Record Dates: First submitted 2016-06-06; First posted 2016-10-12 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Hematological Malignancies
Keywords: Diffuse large B-cell lymphoma (DLBCL); Follicular lymphoma (FL); Mantle cell lymphoma (MCL); Hodgkin lymphoma (HL); Chronic lymphocytic leukemia/small lymphocytic lymphoma; Multiple myeloma (MM); Acute lymphoblastic leukemia (ALL); Acute myeloid leukemia (AML)
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — CBLC137

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBL0137 Dose Escalation (Experimental): * Dose Level 1: 150mg/m2, IV
  * Dose Level 2: 180mg/m2, IV
  * Dose Level 3: 240mg/m2, IV
  * Dose Level 4: 320mg/m2, IV
  * Dose Level 5: 400mg/m2, IV
  * Dose Level 6: 540mg/m2, IV
  * Dose Level 7: 650mg/m2, IV
  * Dose Level 8: 780mg/m2, IV
  * Dose Level 9: 950mg/m2, IV
  * Dose Level 10: 1150mg/m2, IV
  * Dose Level 11: 1400mg/m2, IV
  * Dose Level 12: 1700mg/m2, IV
  * Dose Level 13: 2000mg/m2, IV
  * Dose Level 14: 2400mg/m2, IV
  * Dose Level 15: 2900mg/m2, IV
  * Dose Level 16: 3500mg/m2, IV
  Interventions: Drug: CBL0137

INTERVENTIONS:
Drug: CBL0137 — CBL0137 administered IV weekly on Days 1 and 8 of repeated 21 day treatment cycles. Number of Cycles: 2 or until progression or unacceptable toxicity develops
  Other Names: Curaxin

SUMMARY:
This clinical trial is a Phase 1, open-label, sequential-group, dose-escalation (Part 1) and cohort-expansion study (Part 2) evaluating the safety, pharmacokinetics, pharmacodynamics, and antitumor activity of intravenously (IV) administered CBL0137 in participants with previously treated hematological malignancies.

DETAILED DESCRIPTION:
Part 1 of the study will evaluate the safety and pharmacology of a range of CBL0137 doses administered IV in participants with previously treated lymphomas, including diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), mantle cell lymphoma (MCL), Hodgkin lymphoma (HL), chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), or multiple myeloma (MM). Cohorts of 3 to 6 subjects will be sequentially enrolled at progressively higher dose levels of CBL0137 using a standard 3+3 dose-escalation design. An additional 6 participants may be accrued at the maximum tolerated dose (MTD) or at the recommended dose (RD) to confirm CBL0137 safety and pharmacology as a prelude to further clinical evaluation.

Part 2 of the study provides cohort expansion to further explore the safety, pharmacology, and clinical activity of CBL0137 monotherapy in participants with specific previously treated hematological cancers, including DLBCL, FL, MCL, HL, CLL/SLL, acute lymphoblastic leukemia (ALL), acute myeloid leukemia (AML), and MM. Twelve evaluable participants with each disease type may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an active hematological malignancy:

  * Part 1 (Dose Escalation): Diagnosis of B-cell DLBCL, FL, MCL, HL, CLL/SLL, or MM as documented by medical records.
  * Part 2 (Cohort Expansion): Diagnosis of DLBCL, FL, MCL, HL, CLL/SLL, ALL, MM, or AML as documented in medical records.
* Requirement for therapy of the hematological malignancy due to disease-related symptoms, lymphadenopathy, organomegaly, extranodal organ involvement, or progressive disease.
* Hematological malignancy has been previously treated, has relapsed after or progressed during prior therapy, and has limited potential for benefit from currently available therapy, including hematopoietic stem cell transplantation.
* Presence of measurable disease:

  * For subjects with DLBCL, FL, MCL, HL, or CLL/SLL: presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy (defined as the presence of ≥1 lesion that measures ≥2.0 cm in the longest dimension and ≥1.0 cm in the longest perpendicular dimension as assessed by computed tomography).
  * For subjects with MM, measurable disease with serum monoclonal immunoglobulin protein (M-protein) ≥1 g/dL, or urine M-protein protein ≥200 mg/24 hours, or involved serum free light chain ≥10 mg/dL.
  * For subjects with ALL or AML, presence of >5% blasts in the bone marrow (based on a bone marrow aspirate/biopsy sample with ≥200 nucleated cells and the presence of bone marrow spicules) and/or >1 x 109/L blasts in the peripheral blood (with the restriction that peripheral blast count in subjects with AML must be <50 x 109/L prior to the start of study therapy).
* Completion of all previous therapy (including surgery, radiotherapy, chemotherapy, immunotherapy, or investigational therapy) for the treatment of cancer ≥2 weeks before the start of study therapy. Note: For subjects with AML, the use of hydroxyurea for management of leukocytosis is allowed in Cycle 1 if hydroxyurea is started prior to the initiation of study therapy.

Exclusion Criteria:

* Part 2 (Cohort Expansion): History of another malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin; adequately treated carcinoma in situ without evidence of disease; adequately treated, papillary, noninvasive bladder cancer; other adequately treated Stage 1 or 2 cancers currently in complete remission; or any other cancer that has been in complete remission for ≥2 years.
* Rapidly progressive, clinically unstable central nervous system hematological malignancy. Note: Central nervous system evaluation is only required in subjects with known or suspected central nervous system malignancy.
* Significant cardiovascular disease, including myocardial infarction, arterial thromboembolism, or cerebrovascular thromboembolism, within 6 months prior to start of study therapy; symptomatic dysrhythmias or unstable dysrhythmias requiring medical therapy; angina requiring therapy; symptomatic peripheral vascular disease; New York Heart Association Class 3 or 4 congestive heart failure; uncontrolled Grade ≥3 hypertension (diastolic blood pressure ≥100 mmHg or systolic blood pressure ≥160 mmHg) despite antihypertensive therapy; or history of congenital prolonged QT syndrome.
* Significant screening ECG abnormalities, including unstable cardiac arrhythmia requiring medication, atrial fibrillation/flutter, left bundle-branch block, 2nd-degree atrioventricular (AV) block type II, 3rd degree AV block, Grade ≥2 bradycardia, or QT corrected for heart rate (QTc) >450 msec (for men) or >470 msec (for women).
* Ongoing risk for bleeding due to active gastrointestinal disease or bleeding diathesis.
* Evidence of an ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infections) at the time of start of study therapy. Note: Subjects with localized fungal infections of skin or nails are eligible.
* In subjects with prior progenitor cell transplantation, evidence of ongoing graft-versus-host disease.

Please speak with Investigator for the complete Inclusion/Exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Part 1: Maximum Tolerated Dose (MTD) and Recommended Dose (RD) | At the end of Cycle 1 (each cycle is 21 days)
  MTD is defined as dose level at which ≥6 subjects have been treated and which is associated with a first-cycle dose-limiting toxicity (DLT) in ≤17% of the participants. RD may be the MTD or may be a lower dose within the tolerable dose range. Selection of the RD will be based on consideration of short- and long-term safety information together with available pharmacokinetic, pharmacodynamic, and efficacy data.
Part 2: Overall Response Rate (ORR) | Through study completion, an average of 1 year
  ORR is defined as the proportion of subjects who achieve a complete response (CR), complete response with incomplete blood count recovery (CRi), or partial response (PR) for those with DLBCL, FL, MCL, HL, or CLL/SLL; the proportion of subjects who achieve a CR, CRi, or unconfirmed CR (CRu) for those with ALL; the portion of subjects who achieve a CR or CRi for those with AML; and the proportion of subjects who achieve a stringent CR (sCR), CR, very good PR (VGPR), or PR for those with MM. An ORR of ≥20% is considered the minimum value of potential interest in each of the selected indications.

CONTACTS AND LOCATIONS:
Overall Officials: Langdon Miller, MD, Study Director — CBLI on behalf of Incuron, Inc.
Locations (4):
- United States (4):
  - The Oncology Institute of Hope & Innovation, Whittier, California
  - Claude Sportes, Augusta, Georgia
  - Roswell Park Cancer Institute, Buffalo, New York
  - University Hospitals Case Medical, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No